CLINICAL TRIAL: NCT00842166
Title: Surveillance of Summer Febrile Syndromes of Viral Origin in South of France
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2008 19; 2008-A00793-52
Record Dates: First submitted 2009-02-11; First posted 2009-02-12 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Summer Febrile Syndromes of Viral Origin
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: BLOOD DRAW — specific interview, sequential blood collection to allow virus isolation, molecular and serological diagnostics in patients

SUMMARY:
The aim is to document viral etiologies of isolated fevers and inlfuenza-like syndromes during summertime in South of France in order to better understand the role of known vector-borne viruses such as Toscana virus, West Nile virus during seasonal activity of the arthropod vector. In each of the four cities, a network of general practitioners will be associated in the project to recruit patients who are not hospitalized. The combined involvement of infectious disease specialists and general practitioner will augment the range of patients (mild disease and sever cases) in the study.

ELIGIBILITY:
Inclusion Criteria:

* Old: equal to or higher than 5 years Living in the south of France, without voyage abroad in the 2 weeks preceding inclusion Presenting a fever or a syndrome pseudogripal since less than 7 days without diagnostic orientation nor infectious pathology of body,
* Affiliated with a mode of social security
* After obtaining free and informed of the written assent

Exclusion Criteria:

* Subject whose adhesion with the protocol is improbable according to the investigator
* Expectant mother
* Subject taking part in another clinical trial or in period of exclusion of a preceding clinical trial infectious
* Pathology of body requiring a specific treatment
* Discovered after inclusion d' a pregnancy

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2009-02; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
to document viral etiologies of isolated fevers and inlfuenza-like syndromes during summertime in South of France | 3 years

SECONDARY OUTCOMES:
Identification and characterization of emergent viruses responsible for estival fever in the south of France | 3years

CONTACTS AND LOCATIONS:
Overall Officials: REMI CHARREL, Principal Investigator — Assistance Publique Hopitaux De Marseille
Locations (1):
- Service des Maladies Infectieuses et Tropicales de l'Hôpital Nord, AP-HM, Marseille, France